CLINICAL TRIAL: NCT04775186
Title: Laparoscopic Burch Colposuspension Versus Midurethral Sling for Treatment of Female Stress Urinary Incontinence a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Aliaboeihayagan Ali Mohammed, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: female stress incontinence
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Treatment of Female Stress Urinary Incontinence
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Burch colposuspension (Experimental)
  Interventions: Procedure: Laparoscopic Burch colposuspension and Mid-urethral slings (TVT and TOT)
- midurethral sling (Experimental)
  Interventions: Procedure: Laparoscopic Burch colposuspension and Mid-urethral slings (TVT and TOT)

INTERVENTIONS:
Procedure: Laparoscopic Burch colposuspension and Mid-urethral slings (TVT and TOT) — Laparoscopic Burch colposuspension and Mid-urethral slings (TVT and TOT)

SUMMARY:
To compare the laparoscopic Burch colposuspension with the midurethral slings (TVT, TOT) for treatment of female stress urinary incontinence as regard efficacy and safety.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is defined by the International Continence Society (ICS) as an involuntary loss of urine on physical exertion, sneezing, or coughing (1). It occurs primarily in multiparous women (2).

The prevalence of UI among Egyptian women is high (55%). Aging, low educational level, menopause, higher parity (>3), vaginal delivery, and previous multiple abortions (>3) are significant risk factors for UI(3) Mid-urethral slings (TVT and TOT) are now the recognized worldwide standard of care for the surgical treatment of stress urinary incontinence(4) (5) Mid-Urethral Slings have a very high satisfaction rate (85-90 %) (4) (6), with durability of satisfaction recently demonstrated out to 5-years (79-85 %) as well as a modest 5-year treatment success (43-51 %) (4, 7) Burch colposuspension is a well-accepted technique for surgical management of stress urinary incontinence (SUI), especially when it is associated with urethral hypermobility. it first description in 1961 (8) (9) Originally performed as an open surgical procedure and then Over time, Burch colposuspension has been adapted for laparoscopy, it was long considered as the "gold standard" for the treatment of SUI before emergent of midurethral slings (9) The cure rates for laparoscopic colposuspention is as high as 68.9% to 88.0% whereas recurrence rates remain low, however, it has been reported that the cure rate of retropubic suspension techniques in general decreases steadily from 90% at 1 year to about70% by 10 years postoperatively. After a decline, it seems to reach a plateau at 65-70% at a 20 year follow-up (9) After the Food and Drug Administration (FDA) issued a warning about the use of transvaginal meshes for pelvic organ prolapse (POP) in 2011, there has been much debate about the use of mesh in the MUS continence procedures. Concern is increasing that the use of transvaginal mesh devices to treat SUI and POP have exposed women to avoidable harms following complications such as infection, tissue extrusion, mesh exposure ,mesh shrinkage, and side effects such as severe pain, sexual dysfunction, and repeat surgical interventions (5).

ELIGIBILITY:
Inclusion Criteria:

* 1- All Adult Female patients complaining of stress urinary incontinence attending the voiding dysfunction clinic at Asyut Urology and Nephrology hospital and willing to participate in the study.

Exclusion Criteria:

* 1- Recurrent SUI. 2- Significance Pelvic organ prolapse requiring surgical intervention. 3- Associated Neurologic disorders affecting the lower urinary tract e.g diabetes, spinal cord injury and others.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
● the result of cough stress test. The outcome will be binary: either negative test meaning no leakage at all or positive meaning there is any sort of leakage on stress. The secondary outcome measures will be the scores | 1 year
  ● Accordingly. the patients will be classified into three groups:
  1. Cured: patients who have negative cough stress test and the patient scores 0 on UDI-6.
  2. Improved: patients who have more than 50% improvement in symptoms as determined by UDI-6.
  3. Failed treatment: patients who have less than 50% improvement in symptoms.